CLINICAL TRIAL: NCT03863184
Title: A Multiple-center Phase 2 Study of Acalabrutinib-Lenalidomide-Rituximab (ALR) With an Expansion Cohort of Acalabrutinib-Lenalidomide-Obinutuzumab (ALO) in Patients With Previous Untreated Mantle Cell Lymphoma
Brief Title: Acalabrutinib-Lenalidomide-Rituximab in Patients With Untreated MCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AstraZeneca (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1807019439
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: MRD; Minimal-residual-disease; Treatment naive; Untreated; Frontline; Acalabrutinib; Lenalidomide; Rituximab; Obinutuzumab
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Neoplasm, Residual | interventions — acalabrutinib; Lenalidomide; Rituximab; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Study intervention begins with an induction phase consisting of 12 cycles of acalabrutinib, lenalidomide, and rituximab (ALR). Responding subjects will be eligible to enter a maintenance phase. Subjects will continue maintenance ALR until disease progression, development of unacceptable toxicity, or voluntary withdrawal. Subjects in CR wishing to attempt stem cell collection following at least 6 months of induction treatment can hold lenalidomide for up to 30 days, and restart following stem cell collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALR in Combination (Experimental): Acalabrutinib, lenalidomide, and rituximab in combination
  Interventions: Drug: Acalabrutinib; Drug: Lenalidomide; Drug: Rituximab
- ALO in Combination (Experimental): Acalabrutinib, lenalidomide and obinutuzumab in combination
  Interventions: Drug: Acalabrutinib; Drug: Lenalidomide; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib, oral, 100 mg BID, continuous
  Other Names: CALQUENCE; ACP-196
Drug: Lenalidomide — Lenalidomide, 15 mg for cycle 1, then escalated as tolerated to 20 mg, QD, Days 1-21 out of 28 day cycles
  Other Names: Revlimid
Drug: Rituximab — Rituximab, IV, weekly during Cycle 1, and every other cycle starting with Cycle 4
  Other Names: Rituxan
  Arms: ALR in Combination
Drug: Obinutuzumab — Obinutuzumab on days 1, 8, 15 of cycle 1, day 1 of cycles 2-6, then every 2 cycles
  Other Names: Gazyva
  Arms: ALO in Combination

SUMMARY:
This is a multi-arm phase 2 study to evaluate the preliminary evidence of efficacy and safety of the combination of acalabrutinib, lenalidomide and rituximab (ALR) and acalabrutinib, lenalidomide and obinutuzumab (ALO) in previously untreated mantle cell lymphoma. The study includes an induction phase consisting of 12 cycles of ALR or ALO. Responding subjects will be eligible to enter a maintenance phase. Subjects will continue maintenance ALR or ALO until disease progression, development of unacceptable toxicity, or voluntary withdrawal. Subjects will be followed after completing study intervention every 6 months for alternate anti-cancer therapy and survival.

DETAILED DESCRIPTION:
This is a multi-arm phase 2 study to evaluate the preliminary evidence of efficacy and safety of the combination of acalabrutinib, lenalidomide and rituximab (ALR) and an expansion cohort of acalabrutinib, lenalidomide and obinutuzumab (ALO) in previously untreated mantle cell lymphoma.

The study includes an induction phase consisting of 12 cycles of ALR or ALO. Responding subjects will be eligible to enter a maintenance phase. Subjects will continue maintenance ALR or ALO until disease progression, development of unacceptable toxicity, or voluntary withdrawal. Subjects in complete response wishing to attempt stem cell collection following at least 6 months of induction treatment can hold lenalidomide for up to 30 days, and restart following stem cell collection.

Subjects will be monitored for Minimal Residual Disease (MRD) status in peripheral blood at baseline and completion of 12 cycles of induction treatment using Adaptive Biotechnology Clonoseq assay, and then every 4 cycles.

Subjects will be followed after completing study intervention every 6 months for alternate anti-cancer therapy and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mantle cell lymphoma
* Age ≥ 18 years
* No prior systemic therapy for lymphoma
* Measurable disease defined by a tumor mass ≥ 1.5 cm in one dimension and measurable in two dimensions; measurable spleen disease is allowed
* Treatment should be indicated according to the treating physician
* ECOG performance status ≤ 2
* Required initial laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
  * Platelet count ≥ 75,000 cells/mm3
  * Calculated creatinine clearance ≥ 30 ml/min by Cockcroft-Gault formula
  * Total bilirubin ≤ 2.0 x ULN
  * AST/SGOT and ALT/SGPT ≤ 3.0 x ULN
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use low molecular weight heparin).
* All subjects must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS®.
* Patients of reproductive potential agree to use birth control throughout their participation in this study, and for 28 days following study termination.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days). FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before and continue for at least 28 days after the last dose of lenalidomide (or 2 days after the last dose of acalabrutinib, whichever is longer). FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual activity with a FCBP through one week post last dose even if they have had a successful vasectomy. Men must also agree to refrain from sperm donation during the same timeframe. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Understand and voluntarily sign an ICF prior to any study related assessments and procedures are conducted.
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Patients with blastoid histology
* Patients with known or suspected CNS involvement
* Viral infection with HIV or hepatitis type B or C. Seropositive HBV patients are eligible if they are negative for HBV DNA by PCR and receive concomitant antiviral therapy during treatment and for additional six months after coming off study.
* Prior history of malignancies other than MCL unless the patient has been disease free for ≥ 5 years from the signing of the ICF. Exceptions include basal cell carcinoma or squamous cell carcinoma of the skin; carcinoma in situ of cervix; carcinoma in situ of breast, or localized prostate cancer
* Active uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease).
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer. Patients on moderate CYP3A inhibitors can be considered for study after a washout period of at least 7 days.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.
* Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
* Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
* Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Patients with a history of toxic epidermal necrolysis or Stevens-Johnson syndrome
* Patients that are pregnant or breast feeding
* Known hypersensitivity to any study drug or excipients
* Patient on corticosteroids within two weeks prior to study entry, except for prednisone ≤ 20 mg/day or equivalent for purposes other than treating MCL
* Use of any other experimental drug or therapy within 28 days of baseline
* Patient at high risk for deep vein thrombosis not willing to take DVT prophylaxis
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Known prior exposure to BTK inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Ruan, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan J, Bond DA, Shah BD, Allan JN, Rutherford SC, Gribbin C, Chen Z, Bhinder B, Tam W, Rossi D, Xiang JZ, Hobbie B, Harbhajan M, Sahni TK, Chen GZ, Sigouros M, Inghirami GG, Chen-Kiang S, Elemento O, Maddocks KJ, Leonard JP, Martin P. MRD-driven Initial Therapy of Acalabrutinib and Lenalidomide plus Rituximab (ALR) or Obinutuzumab (ALO) for Mantle Cell Lymphoma. Blood Adv. 2025 Nov 25:bloodadvances.2025017760. doi: 10.1182/bloodadvances.2025017760. Online ahead of print. PMID 41289154
- See also: WCM Joint Clinical Trials Office — https://jcto.weill.cornell.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 patients were consented and 34 were enrolled, with 3 patient deemed as screen failure.
Groups:
- ALR -Cohort A: Patients in Cohort A-ALR will receive combination therapy of acalabrutinib, lenalidomide, and rituximab.
- Cohort B-ALO: Subjects in ALO cohort will get a combination of acalabrutinib, lenalidomide and obinutuzumab
Period: Overall Study
Arm/Group | ALR -Cohort A | Cohort B-ALO
Started | 24 | 10
Completed | 24 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ALO in Combination: Acalabrutinib, Lenalidomide and Obinutuzumab in combination
  Acalabrutinib 100 mg BID continuous
  Lenalidomide on days 1-21 (15 mg for cycle 1, then escalate as tolerated to 20 mg)
  Obinutuzumab on days 1, 8, 15 of cycle 1, day 1 of cycles 2-6, then every 2 cycles
- Total: Total of all reporting groups
Arm/Group | ALR in Combination | ALO in Combination | Total
Number analyzed (Participants) | 24 | 10 | 34
Age, Continuous [Median (Full Range); unit: Years] | 64 [35 to 77] | 65 [37 to 82] | 65 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 19 | 8 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 22 | 8 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Blood Minimum Residual Disease (MRD)-Negative Complete Response (CR) Rate of the Combination of Acalabrutinib + Lenalidomide + Rituximab at the Conclusion of 12 Cycles of Induction Therapy
Description: Percentage of subjects with MRD-negative CR at the conclusion of 12 cycles of induction therapy. Each cycle is 28 days, 12 cycles is approximately 1 year.
Time Frame: 1 year
Population: MRD < 10-6 after 12 cycle induction
Measure: Count of Participants; unit: Participants
Arm/Group | ALR in Combination | ALO in Combination
Number analyzed (Participants) | 24 | 10
Participants | 16 | 9

2. Secondary Outcome: Safety of Combination Treatment With Acalabrutinib, Lenalidomide, and Rituximab as Measured by the Percentage of Subjects That Experience 1 or More Adverse Event
Description: Rate of subjects that experience 1 or more adverse events
Time Frame: 4 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Response Rate
Description: Rate of subjects who achieve a partial or complete response
Time Frame: 4 years
Reporting Status: Not Posted

4. Secondary Outcome: Complete Response Rate
Description: Rate of subjects who achieve a complete response
Time Frame: 4 years
Reporting Status: Not Posted

5. Secondary Outcome: Progression Free Survival
Description: Measured from start of treatment to time of progression or death from any cause, measured in months
Time Frame: 4 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: Measured from start of treatment to death from any cause, measured in months
Time Frame: 4 years
Reporting Status: Not Posted

7. Secondary Outcome: Time to Next Treatment
Description: Measured from end of study treatment to initiation of next lymphoma treatment, measured in months
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AEs will be reported until 30 days after the last dose of study treatment or the start of new anticancer therapy, an average of 2 years.
Arm/Group | ALR -Cohort A | Cohort B-ALO
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/10
Serious Adverse Events (participants affected / at risk) | 16/24 | 4/10
Other Adverse Events (participants affected / at risk) | 24/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALR -Cohort A (N=24) | Cohort B-ALO (N=10)
Fever (General disorders) | 3 (7) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 Infection (Infections and infestations) | 4 (5) | 0 (0)
Lenalidomide Overdose (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Actinic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transverse Myelitis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-related Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALR -Cohort A (N=24) | Cohort B-ALO (N=10)
Anemia (Blood and lymphatic system disorders) | 8 (13) | 3 (12)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 17 (28) | 8 (24)
Platelet count decreased (Investigations) | 7 (8) | 5 (9)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Unspecified tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Hemotypmanum (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Euthyroid Sick Syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyerparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 5 (7) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (3)
Atherosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Coronary Artery Calcification (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (7)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)
Libido decreased (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Creatinine clearance decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Difficult urinating (Renal and urinary disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (6) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac catheterization (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel procedure (Surgical and medical procedures) | 1 (2) | 0 (0)
Cataract surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Dental Procedure, Unspecified (Surgical and medical procedures) | 3 (3) | 0 (0)
Eye sugery (Surgical and medical procedures) | 1 (2) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Laser lithotripsy (Surgical and medical procedures) | 1 (1) | 0 (0)
Moh's procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Mole removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Root canal (Surgical and medical procedures) | 3 (3) | 0 (0)
Scalp cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin lesion removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Skim removal procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (7) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 15 (17) | 9 (12)
Hermitte's Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (3)
Peripheral neuropathy (Nervous system disorders) | 6 (6) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Spacsticity (Nervous system disorders) | 1 (1) | 0 (0)
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Weakness (Nervous system disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye strain (Eye disorders) | 0 (0) | 1 (1)
Stye (Eye disorders) | 1 (2) | 0 (0)
Vision decreased (Eye disorders) | 1 (1) | 0 (0)
Vision disturbance (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 2 (2)
Alopecia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (4) | 4 (4)
Diaphoresis (General disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (3) | 0 (0)
Edema limbs (General disorders) | 5 (6) | 0 (0)
Fatigue (General disorders) | 18 (25) | 5 (7)
Fever (General disorders) | 8 (9) | 4 (5)
Flu-like symptoms (General disorders) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Hair thinning (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 11 (12) | 1 (1)
Irritability (General disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1)
Lymphadenopathy (General disorders) | 1 (1) | 0 (0)
Night sweats (General disorders) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
General pain (General disorders) | 0 (0) | 3 (6)
Pedal Edema (General disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (21) | 5 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (7)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Recurrent organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (11) | 3 (3)
Anal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Burning sensation of tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (14) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 17 (29) | 9 (25)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (14) | 7 (12)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral thrush (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tubular adenoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (6)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 4 (4) | 3 (3)
Transaminitis (Investigations) | 3 (3) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (9) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
LDH increased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6) | 4 (7)
Aspartate aminotransferase increased (Gastrointestinal disorders) | 3 (4) | 4 (9)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (10)
Blood bilirubin increased (Investigations) | 1 (7) | 4 (5)
Creatinine increased (Investigations) | 4 (4) | 3 (5)
INR increased (Investigations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
TSH Elevated (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 8 (10) | 4 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (13) | 3 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (25) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Submandibular tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COVID-19 Infection (Infections and infestations) | 18 (28) | 3 (3)
Yeast infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (6) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (6) | 4 (7)
Shingles (Infections and infestations) | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 2 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Tooth infection (Infections and infestations) | 3 (4) | 1 (1)
Infective rhinitis (Infections and infestations) | 1 (2) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 1 (3)
Herpes infection (Infections and infestations) | 1 (2) | 0 (0)
Viral hepatitis (Infections and infestations) | 1 (1) | 0 (0)
E.coli infection (Infections and infestations) | 0 (0) | 2 (2)
C. difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (2) | 0 (0)
H. pylori infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Head contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Abrasions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Brittle nails (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lipoma (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Molluscum - Right Forearm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Acral nevus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 (43) | 6 (11)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scalp rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrheic Keratitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arcochordons (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Benign cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Precancerous skin scaling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stomach lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03863184/Prot_SAP_000.pdf